CLINICAL TRIAL: NCT05878444
Title: Evaluate the Colonization Capacity of a New Generation Probiotic Within the Project: Valorization of an Intestinal Bacterium as a Functional Ingredient to Prevent the Development of Metabolic Syndrome and Diabetes -BIOPRED
Brief Title: Evaluation of the Colonization Capacity of a Probiotic Bacterium.
Acronym: BIOPRED
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valencian Innovation Agency (Other Government)
Responsible Party: Principal Investigator, Yolanda Sanz Herranz, Full Professor, Institute of Agrochemistry and Food Technology, National Research Council
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INNVA1/2021/32
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Obese; Weight, Body
Keywords: probiotic; Obese; Colonization; Microbiota
MeSH Terms: conditions — Obesity; Body Weight | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: We will try the probiotic in normal weight and overweight/obese people
Who Masked: Outcomes Assessor
Masking Description: Samples will be coded and they will not know the pacient personal/sociodemographic data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight (Experimental): People with BMI between 20-25 will be enrolled in this group. They will take the probiotic capsule daily during 15 days. Dosis will be 10^9-10.
  Interventions: Dietary Supplement: Probiotic
- Overweight/Obese (Experimental): People with BMI >25 will be enrolled in this group. They will take the probiotic capsule daily during 15 days. Dosis will be 10^9-10.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Resistant gastrointestinal capsules will be provided daily to the participants.

SUMMARY:
The goal of this interventional study is to test the colonization of a new generation probiotic in normal weight and overweight/obese people.

The main question aims to answer is if our bacteria is able to colonize the human intestine.

Participants will recieve a probiotic pill every day during 15 consecutive days and fill in questionaries.

DETAILED DESCRIPTION:
Normal weight and overweight volunteers will be recruited to evaluate the colonization capacity of the bacteria. In this case, stool samples will be taken before starting the intervention (T0), after the treatment (T1) and a week after fiinishing the administration of the probiotic (T2). All the subjects will receive the probiotic supplement in capsules taken daily, 7-8 normal weight subjects will take a concentration of 10^9-10 CFU and 7-8 overweight subjects will take a concentration of 10^9-10 CFU.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Body mass index between 20-25 kg/m2 for normopese subjects and BMI 25-30 kg/m2 for overweight participants.
* Body weight and eating habits stable in the last three months before the first visit.
* Willingness to participate in the intervention study, giving their data and samples.
* Signature and acceptance of the informed consent.

Exclusion Criteria:

* Preexistence of other physical conditions (food allergy/sensitivity, gastrointestinal conditions [such as inflammatory bowel disease, celiac disease, pancreatitis, chronic constipation, etc.], immunodeficiency)
* Eating disorders
* Use of antibiotics one month prior to the first visit
* Chronic use of medications (antacids, antidiabetics, anti-hypertensives, etc.)
* History or current abuse of drugs or alcohol
* Following a vegetarian, vegan, or other restrictive diet
* Any other reason deemed appropriate for exclusion at the clinician's discretion
* Non-compliance with adherence to treatment regimen
* Direct association with research and/or investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Presence of our bacteria in feces | Before the end of 2023
  By specific PCR or by 16s sequencing

SECONDARY OUTCOMES:
Adverse effect | Before the end of 2023
  Check if the probiotic is well tolerated. We will collect gastrointestinal symptoms and bristol scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Agrochemistry and Food Technology, Paterna, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
confidentiality and protection of personal data law